CLINICAL TRIAL: NCT01543347
Title: Temocillin Use in Complicated Urinary Tract Infections Due to Extended Spectrum Beta-Lactamases (ESBL) Producing and AmpC Hyperproducing Enterobacteriaceae in United Kingdom
Brief Title: Temocillin Use in Complicated Urinary Tract Infections Due to Extended Spectrum Beta-Lactamases (ESBL)/AmpC Enterobacteriaceae
Acronym: TEA
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No patient has been included in 9 months because of strict incl/excl criteria
Sponsor: Belpharma s.a. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMO-07001; 2008-005912-41 (EudraCT Number)
Record Dates: First submitted 2012-02-22; First posted 2012-03-05 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Urinary Tract Infection
Keywords: UTI; ESBL; AmpC Enterobacteriaceae
MeSH Terms: conditions — Urinary Tract Infections | interventions — temocillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temocillin (Experimental): Treatment group
  Interventions: Drug: Temocillin

INTERVENTIONS:
Drug: Temocillin — Antibiotic treatment
  Other Names: Negaban

SUMMARY:
This study is aimed at demonstrating the efficacy of temocillin in the treatment of complicated Urinary Tract Infection (UTI) due to confirmed Extended Spectrum Beta-Lactamases (ESBL) producing or AmpC hyperproducing Enterobacteriaceae in the United Kingdom.

DETAILED DESCRIPTION:
The spectrum of activity together with the route of excretion of temocillin makes it a good candidate for the treatment of urinary tract infections. Several studies have shown very good clinical and microbiological activity in uncomplicated and complicated cystitis and pyelonephritis in adults and in pyelonephritis in children older than 2 months. However there is no specific study performed on Urinary Tract Infections due to broad spectrum ß-lactamases producing strains.

In this context, this study is aimed at demonstrating the efficacy of temocillin in the treatment of complicated Urinary Tract Infection due to confirmed Extended Spectrum Beta-Lactamases (ESBL) producing or AmpC hyperproducing Enterobacteriaceae in the United Kingdom. The investigators will also evaluate the tolerance of the drug by monitoring the adverse event and the incidence of eventual Clostridium difficile associated infection.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting a complicated urinary tract infection due to a confirmed Extended Spectrum Beta-Lactamases (ESBL) producing or AmpC hyperproducing Enterobacteriaceae susceptible to temocillin requiring parenteral antimicrobial therapy.
* community or hospital acquired infecting bacteria.
* signed informed consent

Exclusion Criteria:

* patients infected with a strain resistant to temocillin
* patients having received an active antimicrobial therapy during the 48h before the beginning of temocillin treatment except temocillin
* patients presenting another site of infection than urinary (except onset of bacteremia from urinary tract origin) due to Gram negative bacteria
* patients needing concomitant antimicrobial therapy with the exception of benzylpenicillin
* uncomplicated cystitis
* complete obstruction of the urinary tract
* prostatitis
* peri-nephretic or intrarenal abscesses
* renal transplant
* children (up to 18 years old)
* pregnancy or lactation
* chronically dialyzed patients
* immunocompromising therapy or illness
* known allergy to penicillin

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Microbiological cure | End of treatment (minimum 5 days)
  Eradication : < 10,000 Colony forming Unit/mL (CFU/mL) of the baseline pathogen
  * Persistence : = 10,000 CFU/mL of the baseline pathogen
  * Persistence with acquisition of resistance
  * Superinfection : = 100,000 CFU/mL of another uropathogen during therapy
  * New infection : = 100,000 CFU/mL of another uropathogen after therapy
  * Relapse : eradication at end of treatment but = 10,000 CFU/mL of the baseline pathogen at follow up
  * Relapse with acquisition of resistance

SECONDARY OUTCOMES:
Clinical cure | End of treatment (minimum 5 days)
  Clinical status of the patient will be classified as
  * cured (resolution of all clinical symptoms)
  * improved
  * failure (persistence of baseline clinical symptoms or emergence of new symptoms)
Development of resistance during treatment | End of treatment (minimum 5 days)
  Acquisition of resistance to temocillin during treatment on a microbiological point of view
Infection relapses monitored over 4-6 weeks | End of follow-up (up to 6 weeks)
  * Relapse : eradication at end of treatment but = 10,000 CFU/mL of the baseline pathogen at follow up
  * Relapse with acquisition of resistance
Monitoring of AE | From day 0 to up to 6 weeks
  Record of any untoward medical occurrence in a clinical trial patient administered temocillin and which does not necessarily have to have a causal relationship with the treatment.
ESBL & AmpC fecal carriage (optional) | Start and end of treatment (minimum 5 days)
  All isolates of included patients will be kept frozen at -80°C and sent to the central laboratory for ESBL/AmpC confirmation and typing through molecular techniques. Pulse field gel electrophoresis will be performed on isolates from the same species for determination of clonality.
Incidence of C. difficile infection | From day 0 to up to 6 weeks
  Clostridium difficile infection (CDI) is defined as recommended by the HPA Steering Group on Healthcare Associated Infection 35 : one episode of diarrhoea, defined either as stool loose enough to take the shape of a container used to sample it, or as Bristol Stool Chart types 5-7, which is not attributable to any other cause including medicines which occurs at the same time as a positive toxin assay (with or without a positive C. difficile culture) and/or endoscopic evidence of pseudomembranous colitis.

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Hawkey, Professor, Principal Investigator — Birmingham Public Health Laboratory
Locations (1):
- Birmingham Heartlands Hospital, Birmingham, United Kingdom